A Prospective Cohort Study on Risk Factors for Postoperative Cough in Patients Undergoing Thoracoscopic Lung Resection

Statistical Analysis Plan

Count data are expressed in terms of frequency and percentage (%) and are based on standards Chi-square test for comparisons between different groups; Conforms to a normal distribution The independent samples T-test was used for the continuous data of, and was expressed as mean  $\pm$  standard deviation. Measurement data that do not conform to the normal distribution are used Wilcoxon's rank-sum test, measured as the median and the 25th (Q1), 75 (Q3) quantile representation; Multivariate logistic regression analysis was used to explore the independent risk factors of CAP. Alluvial Diagrams will be used to represent groups over the course of three follow-ups. The Leicester score is used to represent the wave of change in the trajectory of the VAS score Move; Group-based trajectory modeling will be used to represent changes in VAS score trajectories.